CLINICAL TRIAL: NCT03162731
Title: A Pilot Trial of Nivolumab and Ipilimumab in Combination With Radiotherapy in Patients With Locally Advanced Head and Neck Cancer; CA209-931
Brief Title: Nivolumab, Ipilimumab, and Radiation Therapy in Treating Patients With Stage III-IVB Head and Neck Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17P.082; JT 10025 (Other: JeffTrial Number)
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Larynx; Lip, Oral Cavity and Pharynx
MeSH Terms: conditions — Laryngeal Diseases; Lymphoid Interstitial Pneumonia | interventions — Nivolumab; Ipilimumab; CTLA-4 Antigen; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment ( nivolumab, ipilimumab, radiation therapy) (Experimental): Patients receive nivolumab IV over at least 30 minutes every 2 weeks and ipilimumab IV over at least 90 minutes every 6 weeks. Beginning week 3, patients undergo simultaneous integrated boost intensity modulated radiation therapy or volumetric modulated arc therapy for 5 days per week over 7 weeks. Patients continue nivolumab every 2 weeks for 12 doses and ipilimumab every 6 weeks for 4 doses. Courses repeat for up to 23 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab; Biological: Ipilimumab; Radiation: Simultaneous-Integrated Boost Intensity-Modulated Radiation Therapy; Radiation: Volume Modulated Arc Therapy

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: 946414-94-4; BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Biological: Ipilimumab — Given IV
  Other Names: 477202-00-9; 720801; 732442; Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Radiation: Simultaneous-Integrated Boost Intensity-Modulated Radiation Therapy — Undergo simultaneous integrated boost integrated modulated radiation therapy
  Other Names: IMRT-SIB; Intensity Modulated Radiation Therapy Simultaneous Integrated Boost; SIB-IMRT
Radiation: Volume Modulated Arc Therapy — Undergo volumetric modulated arc therapy
  Other Names: VMAT

SUMMARY:
This pilot clinical trial studies the side effects of nivolumab, ipilimumab and radiation therapy in treating patients with stage IVA-B head and neck cancer. Monoclonal antibodies, such as nivolumab and ipilimumab, may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving nivolumab, ipilimumab, and radiation therapy may work better in treating patients with stage IVA-B head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the safety of the combination of nivolumab and ipilimumab with radiation treatment for definitive management of patients with locally advanced squamous cell carcinoma of the head and neck.

SECONDARY OBJECTIVES:

I. To estimate the 1 year progression-free survival (PFS) in all patients treated.

II. To assess the overall response rate and overall survival of patients at one year

TERTIARY OBJECTIVES:

I. To explore whether PDL1 expression is associated with treatment response. II. To explore whether there is a net change in the Th1/Th2 ratio (IFN-gamma, IL-4, IL10, etc) or cell subset frequencies (M2 monocytes, myeloid-derived suppressor cells, etc) within a patient's peripheral blood either at baseline or in response to treatment is associated with treatment response.

III. To explore whether exosomes or other immune related serum biomarkers change after combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age and older
* Pathologically confirmed squamous cell carcinoma of the head and neck (SCCHN), not previously treated
* Stage III-IVB disease of 1) oral cavity, 2) HPV-negative (p16-) oropharynx, 3) larynx, 4) hypopharynx
* Oropharyngeal primaries that are HPV-mediated (p16+) must be stage II-III. Stage II pateints must be either N2 or, if T3N0 or T3N1 they must also have at least 20 pack year history of smoking
* Tumor sample must be available for HPV p16 and PD-L1 testing
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* White blood cells 2000/ul or more
* Absolute neutrophil count 1500/ul or more
* Platelets 100,000/ul or more
* Hemoglobin 9 g/dl or more
* Bilirubin less than or equal to 1.5 x the upper limit of normal (except subjects with Gilbert syndrome, who can have total bilirubin < 3 mg/dl)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x the upper limit of normal
* Glomerular filtration rate (GFR) greater than or equal to 40 ml/min using the Cockcroft-Gault formula or Serum creatinine less than or equal to 1.5 x upper limit of normal (ULN)
* Women of reproductive potential should have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours of the start of study drugs
* Women of reproductive potential must use highly effective contraception methods to avoid pregnancy for 23 weeks after the last dose of study drugs; "women of reproductive potential" is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level more than 40 mIU/mL
* Men of reproductive potential who are sexually active with women of reproductive potential must use any contraceptive method with a failure rate of less than 1% per year; men who are receiving the study medications will be instructed to adhere to contraception for 31 weeks after the last dose of study drugs; men who are azoospermic do not require contraception
* Informed consent: all subjects must be able to comprehend and sign a written informed consent document

Exclusion Criteria:

* Primary nasopharyngeal carcinoma
* Patients with brain metastases
* Patients who have participated in a study with an investigational agent or device within 2 weeks of initiation of treatment
* Any prior radiotherapy to the neck
* Patients with known contraindications to radiotherapy, including inherited syndromes associated with hypersensitivity to ionizing radiation (e.g., Ataxia-Telangiectasia, Nijmegen Breakage Syndrome)
* Any prior chemotherapy or radiation therapy for the current diagnosis
* Any prior therapy with anti-PD-1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Any history of a sever hypersensitivity reaction to any monoclonal antibody
* Any history of allergy to the study drug components
* Any concurrent malignancies- exceptions include- basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer or in situ cervical cancer that has undergone potentially curative therapy; patients with a history of other prior malignancy must have been treated with curative intent and must have remained disease-free for 3 years post-diagnosis
* Any diagnosis of immunodeficiency or current immunosuppressive therapy including >10mg/day of prednisone within 14 days of enrollment is not permitted
* Patients that have an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids (> 10 mg daily prednisone equivalents) or immunosuppressive agents; subjects with vitiligo, type I diabetes mellitus, or resolved childhood asthma/atopy would be an exception to this rule. Inhaled or topical steroids, and adrenal replacement steroids </=10mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study
* Patients with evidence of interstitial lung disease or active, non-infectious pneumonitis
* Patients with a known human immunodeficiency virus infection (HIV 1/2 antibodies) or acquired immunodeficiency syndrome (HIV/AIDS), active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Patients who have received a live vaccine within 30 days prior to the radiation therapy
* Patients must not be receiving any other investigational agents
* Patients with uncontrolled intercurrent illnesses including, but not limited to an active infection requiring systemic therapy or a known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the trial
* Women must not be pregnant (as above) or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2020-09-27 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events assessed using Common Terminology Criteria for Adverse Events version 4.03 | Up to 6 months
  There will be continuous monitoring of the incidence of grade 3-5 toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Johnson, MD, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Johnson JM, Vathiotis IA, Harshyne LA, Ali A, Bar Ad V, Axelrod R, Lorber E, Curry J, Cognetti DM, Luginbuhl AJ, Tuluc M, Keith S, Mahoney MG, Argiris A. Nivolumab and ipilimumab in combination with radiotherapy in patients with high-risk locally advanced squamous cell carcinoma of the head and neck. J Immunother Cancer. 2023 Aug;11(8):e007141. doi: 10.1136/jitc-2023-007141. PMID 37536941
- [Derived] Ali AS, Manukian G, Johnson JM, Vathiotis I, Axelrod R, Keith SW, Curry J, Cognetti D, Luginbuhl A, Argiris A, Bar-Ad V. In-Field Toxicity Analysis of a Phase 1 Clinical Trial of Nivolumab and Ipilimumab With Definitive Radiation Therapy in Locally Advanced Squamous Cell Carcinoma of the Head and Neck. Int J Radiat Oncol Biol Phys. 2023 Sep 1;117(1):181-185. doi: 10.1016/j.ijrobp.2023.03.065. Epub 2023 Apr 3. No abstract available. PMID 37019367
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/